CLINICAL TRIAL: NCT03478280
Title: Effect of Brodalumab Compared to Placebo on Vascular Inflammation in Moderate-to-severe Psoriasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Principal Investigator, Anne Bregnhøj, MD, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PsoPET2
Record Dates: First submitted 2018-03-13; First posted 2018-03-27 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Intervention Model Description: A randomised, double-blind, placebo-controlled, trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brodalumab (Active Comparator): Subjects will receive 210 mg of Kyntheum administered by subcutaneous injection at Weeks 0, 1 and 2 followed by 210 mg every other week (EOW) thereafter.
  Interventions: Drug: Brodalumab
- Placebo (Placebo Comparator): Subjects will receive placebo doses administered by subcutaneous injection at Weeks 0, 1 and 2 followed by placebo EOW thereafter.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Brodalumab — Subjects with moderate-to-severe psoriasis are enrolled consecutively and randomly assigned to either active treatment with brodalumab or placebo during the treatment period
  Other Names: Kyntheum
  Arms: Brodalumab
Drug: Placebos — Subjects with moderate-to-severe psoriasis are enrolled consecutively and randomly assigned to either active treatment with brodalumab or placebo during the treatment period
  Arms: Placebo

SUMMARY:
A randomised, double-blind, placebo-controlled, trial to evaluate the efficacy of brodalumab monotherapy on vascular and systemic inflammation by 18F-FDG-PET/CT in subjects with moderate-to-severe plaque-type psoriasis who are candidates for systemic therapy

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject prior to performing any protocol-related procedures.
2. Age 40 and above.
3. Diagnosis of chronic plaque psoriasis confirmed by a dermatologist
4. PASI ≥ 10

Exclusion Criteria:

1. Non-Danish speaking
2. Known or suspected allergy or reaction to any component of the IMP formulation.
3. History of inflammatory bowel disease, arthritis (not including psoriatic arthritis), systemic lupus erythematosus, and active inflammatory skin diseases.
4. A history of malignancies within the past five years (excluding localized non-melanoma skin cancer).
5. Topical corticosteroid treatment (class III or stronger) and/or ultraviolet type B phototherapy within 2 weeks prior to randomization
6. Treatment with psoralen plus ultraviolet type A photochemotherapy, methotrexate, cyclosporine, acitretin, or fumaric acid esters within 4 weeks prior to randomization.
7. Treatment with adalimumab, etanercept, infliximab, cosentyx, or ixekizumab within 12 weeks, ustekinumab within 24 weeks, or other immunosuppressive or anti-inflammatory agents within 5 half-lives of the active substance prior to the FDG-PET/CT, respectively.
8. Scheduled surgery during the trial period (expect minor minimally invasive procedures).
9. Systemic infection or fever within 7 days prior to FDG-PET/CT.
10. Severe obesity (> 150 kg due to a PET/CT scanner limitation).
11. Presence of uncontrolled diabetes mellitus (HbA1c > 75 mmol/mol and/or blood sugar > 11.1 mmol/l and/or clinical judgment).
12. History of coagulation defects (clinical judgment).
13. Active or latent tuberculosis requiring treatment.
14. Positive hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb), hepatitis B core antibody (HBcAb) or hepatitis C virus antibody (anti-HCV) serology at screening. Subjects with positive HBsAb may be randomised provided they are hepatitis B vaccinated and have negative HBsAg and HBcAb.
15. History of any known primary immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test at screening, or the subject taking antiretroviral medications as determined by medical history and/or subject's verbal report.
16. No history of varicella zoster infection and negative varicella antibody test (until varicella vaccination is completed).
17. History of chronic alcohol or drug abuse within 12 months prior to screening, or any condition associated with poor compliance as judged by the investigator.
18. History of intravenous drug use.
19. History of attempted suicide or is at significant risk of suicide.
20. Major surgery within the past 3 months.
21. Pregnancy or lactation (Women of childbearing potential must use a highly effective* form of birth control (confirmed by the investigator) throughout the trial and until 12 weeks after discontinuation of treatment with brodalumab.
22. Claustrophobia.
23. Reduced renal function (serum creatinine > 200 μmol/L or cr-EDTA clearance < 30 ml/min)
24. Any disorder, including but not limited to, cardiovascular, lung, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, immunological, psychiatric, or major physical impairment that is not stable, in the opinion of the investigator, and could:

    * Affect the safety of the subject throughout the trial.
    * Influence the findings of the trial or their interpretations.
    * Impede the subject's ability to complete the entire duration of trial.

      * A highly effective method of birth control is defined as one which results in a low failure rate (less than 1% per year) such as bilateral tubal occlusion, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), sexual abstinence (when this is in line with the preferred and usual life style of the subject), vasectomised partner (given that the subject is monogamous). The subjects must have used the contraceptive method continuously for at least 1 month prior to the pregnancy test. A female is defined as not being of child bearing potential if she is postmenopausal (at least 12 months with no menses without an alternative medical cause prior to screening), or surgically sterile (hysterectomy, bilateral salpingectomy or bilateral oophorectomy).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
The aortic wall inflammation at baseline and at week 16 in brodalumab treated psoriasis subjects compared to placebo. | 16 weeks
  The average of maximum TBR values (MeanTBRmax) of the entire aorta at baseline and at week 16

SECONDARY OUTCOMES:
The splenic inflammation at baseline and at week 16 in brodalumab treated psoriasis subjects compared to placebo. | 16 weeks
  The spleen-to-liver ratio (SLR) based on splenic and liver mean standardised uptake values (SUVmean)
The aortic wall subsegment inflammation at baseline and at week 16 in brodalumab treated psoriasis subjects compared to placebo. | 16 weeks
  The average of maximum TBR values (MeanTBRmax) of the ascending, aortic arch, descending, suprarenal, and infrarenal aorta at baseline and at week 16
The skin inflammation at baseline and at week 16 in brodalumab treated psoriasis subjects compared to placebo. | 16 weeks
  Severity of psoriasis measured by PASI score at baseline and at week 16

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT03478280/Prot_ICF_000.pdf